CLINICAL TRIAL: NCT05877599
Title: An Open-label, Phase 1, Multicenter Study to Evaluate the Safety and Preliminary Anti-tumor Activity of NT-175 in Human Leukocyte Antigen-A*02:01-Positive Adult Subjects With Unresectable, Advanced and/or Metastatic Solid Tumors That Are Positive for the TP53 R175H Mutation
Brief Title: A Study of NT-175 in Adult Subjects With Unresectable, Advanced, and/or Metastatic Solid Tumors That Are Positive for HLA-A*02:01 and the TP53 R175H Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-175-201
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Carcinoma; Pancreatic Adenocarcinoma; Breast Cancer; Other Solid Tumors; Ovarian Cancer
Keywords: Cell therapy; TP53; Solid tumors; Non-small cell lung cancer; Head and neck squamous cell carcinoma; Colorectal carcinoma; Pancreatic adenocarcinoma; Breast Cancer; Ovarian Cancer; TCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation and Expansion (Experimental): Dose Escalation of TCR T cell product
  Interventions: Biological: Autologous, engineered T Cells targeting TP53 R175H
- Part 1: Disease Histology Evaluation (Experimental): TCR T Cell Product at the MTD
  Interventions: Biological: Autologous, engineered T Cells targeting TP53 R175H
- Part 2: Disease Cohort Expansion (Experimental): TCR T Cell Product at the RP2D
  Interventions: Biological: Autologous, engineered T Cells targeting TP53 R175H

INTERVENTIONS:
Biological: Autologous, engineered T Cells targeting TP53 R175H — * Pre-conditioning by non-myeloablative chemotherapy with fludarabine and cyclophosphamide
  * Single infusion TCR T cells
  * Post-infusion recombinant interleukin-2 (rIL-2)

SUMMARY:
Phase I Study of NT-175, an autologous T cell therapy product genetically engineered to express an HLA-A*02:01-restricted T cell receptor (TCR), targeting TP53 R175H mutant solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter study to evaluate the safety and preliminary antitumor activity of NT-175 in HLA-A*02:01 subjects with unresectable, advanced, and/or metastatic NSCLC, colorectal adenocarcinoma, HNSCC, pancreatic adenocarcinoma, ovarian cancer, breast cancer, or any other solid tumor histologies that are positive for the TP53 R175H mutation.

Dose Escalation will investigate escalating doses of NT-175 in adult subjects with eligible solid tumor histologies and will evaluate the safety and MTD.

Disease Histology Evaluation will further evaluate the safety and preliminary anti-tumor activity at or below the MTD in disease specific histologies and determine the RP2D. .

Disease Cohort Expansion will further evaluate the preliminary anti-tumor activity and safety of NT-175 at the RP2D in disease specific settings.

ELIGIBILITY:
Key Inclusion Criteria

* Subjects must be at least 18 years of age, at the time of signing the informed consent.
* Subjects must be capable of giving signed informed consent.
* Subject must be diagnosed with one of the histologies below:

  * NSCLC
  * Colorectal adenocarcinoma
  * HNSCC
  * Pancreatic adenocarcinoma
  * Breast cancer
  * Ovarian cancer
  * Any other solid tumor
* Tumors must harbor a TP53 R175H variant mutation and subject must be HLA-A*02:01 positive (at least 1 allele) as confirmed by an CLIA-accredited laboratory-based test.
* Subject has advanced solid cancer, defined as unresectable, advanced, and/or metastatic disease (Stage III or IV) after at least 1 line of approved systemic standard of care (SOC) treatment regimen and for which there are no available curative treatment options.
* Subject has at least 1 measurable lesion per computed tomography (CT) scan or magnetic resonance imaging (MRI) per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at the time of enrollment
* Adequate hematological, renal, hepatic, pulmonary, and cardiac function
* Per Investigator judgement, subject is likely to complete study visits and/or procedures per the protocol and comply with study requirements for study participation

Key Exclusion Criteria

* Any another primary malignancy within the 3 years prior to enrollment (except for non-melanoma skin cancer, carcinoma in situ (eg, cervix, bladder, breast) or low-grade prostate cancer
* Known, active primary central nervous system (CNS) malignancy
* History of prior adoptive cell and gene therapy, allogeneic stem cell transplant or solid organ transplantation.
* History of stroke or transient ischemic attack within the 12 months prior to enrollment.
* History of clinically significant cardiac disease within the 6 months prior to enrollment or heart failure at any time prior to enrollment.
* Systemic therapy within at least 2 weeks or 3 half-lives, whichever is shorter, prior to enrollment.
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or rIL-2; or known sensitivity or allergy to methotrexate, gentamicin, or other aminoglycosides.
* Any form of primary immunodeficiency.
* Live vaccine ≤ 4 weeks prior to enrollment or plans to have a live vaccine prior to planned lymphodepleting chemotherapy and/or NT-175 treatment.
* Active immune-mediated disease requiring systemic steroids or other immunosuppressive treatment (except if related to prior checkpoint inhibitor therapy)
* Female of childbearing potential who is lactating or breast feeding at the time of enrollment.
* Known to have Li-Fraumeni syndrome or is known to have relatives who are diagnosed with Li-Fraumeni syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Safety of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | 28 days after infusion
  Incidence of dose-limiting toxicities (DLTs) after the infusion of NT-175
Part 1: Safety of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months post-infusion
  Incidence of adverse events and serious adverse events
Part 2: Further Evaluate the safety of NT-175 at the RP2D in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Treatment-emergent adverse events, and serios adverse events
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Objective Response Rate (ORR) per RECIST V1.1 determined by Investigator assessment.
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Best Overall Response (BOR) per RECIST V1.1 determined by Investigator assessment.
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Duration of Response (DOR) per RECIST V1.1 determined by Investigator assessment.
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Clinical Benefit Rate (CBR) per RECIST V1.1 determined by Investigator assessment.
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Time to Response (TTR) per RECIST V1.1 determined by Investigator assessment.
Part 2: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Progression-free survival (PFS) per RECIST V1.1 determined by Investigator assessment.

SECONDARY OUTCOMES:
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Objective Response Rate (ORR) per RECIST V1.1 determined by Investigator assessment.
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Best Overall Response (BOR) per RECIST V1.1 determined by Investigator assessment.
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Duration of Response (DOR) per RECIST V1.1 determined by Investigator assessment.
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Clinical Benefit Rate (CBR) per RECIST V1.1 determined by Investigator assessment.
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Time to Response (TTR) per RECIST V1.1 determined by Investigator assessment.
Part 1: Preliminary anti-tumor activity of NT-175 in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Progression-free survival (PFS) per RECIST V1.1 determined by Investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca, Study Director — AstraZeneca
Locations (18):
- United States (18):
  - Research Site, Gilbert, Arizona
  - Research Site, Duarte, California
  - Research Site, Newport Beach, California
  - Research Site, Santa Monica, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/